CLINICAL TRIAL: NCT02995564
Title: The Multi-Media Social Skills Project for Adults: Validation of an Intervention for Adults With Autism Spectrum Disorders
Brief Title: The Multi-Media Social Skills Project for Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Pennsylvania Bureau of Autism Services (Other)
Responsible Party: Principal Investigator, Michael Murray, Director of the Division of Autism Services, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41078EP
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Autism Spectrum Disorders
Keywords: Social Skills; Asperger's; High-functioning autism; Young adults
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Social Skills Intervention (Experimental): The intervention is a 16-week social skills therapy program that will consist of a 90 minute group therapy session followed by a 90 minute peer generalization session meeting once per week. Each cohort will consist of 6 adolescents with Aspergers or high-functioning autism, who will be joined by 6 typically-developing peers for the peer generalization portion. During the group therapy session young adults will discuss and watch video clips addressing social skills topics relevant to their age group. They will have a chance to practice these skills when paired with typically developing peer volunteers.
  Interventions: Behavioral: social skills therapy

INTERVENTIONS:
Behavioral: social skills therapy — Sixteen week manual based social skills curriculum targeting social fluency and responsiveness.

SUMMARY:
This study is investigating the development of a social skills training program for adults with Asperger's Syndrome or high-functioning autism, ages 18 to 35 years. The Principal Investigator for this study is Dr. Michael Murray, the director of the Autism Studies Division at the Penn State Hershey Medical Center. The purpose of this study is to adapt a social skills training program to address and enhance the social skills of adults with Asperger's Syndrome and high-functioning autism.

DETAILED DESCRIPTION:
During group study visits, a group of six young adults with Asperger's Syndrome or high-functioning autism will meet weekly for about 90 minutes. The purpose of the group sessions is to work on everyday social skills such as initiating and maintaining conversations, establishing friendships, and dealing with situations such as job interviews and dating.

A generalization session will be held every week after the group therapy session with same-age peers who have been screened to participate in the study. The purpose of including peers in the class is to give young adults with Asperger's syndrome and high-functioning autism a chance to practice the social skills learned in the group study visit with a peer group. Study participants will be paired with a typically developing peer for an outing in the community to a nearby restaurant or shop or an in-class exercise such as a mock job interview.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 35 years of age
* Must be a Pennsylvania resident
* A primary diagnosis of Asperger's Syndrome or high-functioning autism, as confirmed by the SRS-2
* A verbal IQ of 85 or above on the Kaufman Brief Intelligence Test, Second Edition
* English as primary language spoken
* Ability to fluently speak in full sentences

Exclusion Criteria:

* A significant language delay
* Difficulty with aggression directed at peers
* A primary thought disorder
* A secondary disorder of anxiety or depression so severe as to prevent the individual's participation in the treatment
* A current high school student at start of intervention
* Low social motivation demonstrated through formalized assessment and/or by responses given to screening interview

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2013-07; Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Social Responsiveness Scale - Adult | One week post-intervention
  The Social Responsiveness Scale - Adult is used to measure levels of social awareness, cognition, communication, motivation, and autistic mannerisms in adults.
Video recording of Social Interaction | One week post-intervention
  Participants will be filmed in a brief interaction with a typically developing peer which will be coded to obtain social interaction skills and fluency scores.

SECONDARY OUTCOMES:
Achenbach Adult Behavior Checklist | One week post-intervention
  The Achenbach is a 126-item survey that asks about behaviors, problems, and substance use.
Social and Emotional Loneliness Scale for Adults (SELSA) | one week post-intervention
  The SELSA is a 37-item survey that assesses friendships and other relationships.
Social Skills Inventory (SSI) | one week post-intervention
  The SSI is a 90-item survey that measures social competence.
Social Phobia Inventory (SPIN) | one week post-intervention
  The SPIN is a 17-item survey that asks about feelings in social situations.
Empathy Quotient | one week post-intervention
  The EQ is a 60-item survey that assesses ability to relate to others.
Achenbach Adult Behavior Checklist - Self Report | one week post-intervention
  A 126-item survey that asks about behaviors, problems, and substance use.
Social Fluency Assessment | one week post-intervention
  Participants will be filmed in a brief interaction with a typically developing peer. These videos will be analyzed for indicators of social fluency such as eye contact, seconds of silence and number of questions asked.
Achenbach Adult Behavior Checklist | three months post-intervention
  The Achenbach is a 126-item survey that asks about behaviors, problems, and substance use.
Social and Emotional Loneliness Scale for Adults (SELSA) | three months post-intervention
  The SELSA is a 37-item survey that assesses friendships and other relationships.
Social Skills Inventory (SSI) | three months post-intervention
  The SSI is a 90-item survey that measures social competence.
Social Phobia Inventory (SPIN) | three months post-intervention
  The SPIN is a 17-item survey that asks about feelings in social situations.
Empathy Quotient | three months post-intervention
  The EQ is a 60-item survey that assesses ability to relate to others.
Achenbach Adult Behavior Checklist - Self Report | three months post-intervention
  A 126-item survey that asks about behaviors, problems, and substance use.
Social Fluency Assessment | three months post-intervention
  Participants will be filmed in a brief interaction with a typically developing peer. These videos will be analyzed for indicators of social fluency such as eye contact, seconds of silence and number of questions asked.
Social Responsiveness Scale - Adult | three months post-intervention
  The Social Responsiveness Scale - Adult is used to measure levels of social awareness, cognition, communication, motivation, and autistic mannerisms in adults.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Murray, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- The Pennsylvania Psychiatric Institute Northeast Drive Clinic, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No